CLINICAL TRIAL: NCT07108517
Title: A Manualized Post-Traumatic Growth Intervention for People With Cancer in Greece - IC-Growth. The Overarching Aim of IC-Growth is to Promote Psychosocial Care and Support for People With Cancer Using Acceptance and Committment Therapy.
Brief Title: A Manualized Post-Traumatic Growth Intervention for People With Cancer in Greece - IC-Growth
Acronym: IC-Growth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Research and Technology Hellas (Other)
Collaborators: AHEPA University Hospital (Other); Hellenic Cancer Society (Other); Theagenio Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Christina Karamanidou, Health Psychologist, Researcher, PhD, Centre for Research and Technology Hellas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ELIDEK_KARAMANIDOU
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Colon Cancer; Head and Neck Cancers
Keywords: Post-Traumatic Growth (PTG); Cancer Survivorship; Psychosocial Intervention; Acceptance and Commitment Therapy (ACT); Quality of Life (QoL); Biomarkers (Cortisol, CRP); Randomized Controlled Trial (RCT; Oncology Supportive Care; Group Therapy; Breast Cancer; Head and Neck Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Head and Neck Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Group-Based Post-Traumatic Growth (PTG) Intervention (Experimental): Participants receive a manualized, group-based psychosocial intervention designed to enhance post-traumatic growth (PTG). The program is delivered over 6-8 weeks, with weekly 90-minute sessions, and incorporates evidence-based techniques (e.g., Acceptance and Commitment Therapy, mindfulness, cognitive and narrative exercises, and interpersonal support).
  Interventions: Behavioral: IC-Growth ACT-Based Support Program
- 2. Standard Care (Usual Oncology Follow-Up) (No Intervention): Participants receive standard oncology follow-up care with no additional psychosocial intervention. They will complete the same assessments as the intervention group at baseline and post-intervention.

INTERVENTIONS:
Behavioral: IC-Growth ACT-Based Support Program — IC-Growth Psychosocial Group Intervention is a structured, manualized program designed to enhance post-traumatic growth (PTG) in adults diagnosed with breast, colorectal, or head and neck cancer. The intervention is delivered in small groups (8-10 participants) over 6-8 weeks, with weekly 90-minute sessions led by trained health psychologists. The program integrates evidence-based therapeutic approaches, including Acceptance and Commitment Therapy (ACT), mindfulness, cognitive restructuring, narrative exercises, and interpersonal support-building, with the goal of improving psychological flexibility, resilience, quality of life, and overall well-being.
  Other Names: Experimental; 1
  Arms: 1. Group-Based Post-Traumatic Growth (PTG) Intervention

SUMMARY:
Cancer can be a very traumatic experience for the people affected and the majority of the psychological literature focuses on this. Less proliferated and researched is the increasingly recognized fact that as a result of struggling with such traumatic adversities, some people experience what is known as post-traumatic growth (PTG). PTG not only allows them to overcome their trauma (e.g., impact of cancer) and return to pre-diagnosis functioning (e.g., health, wellbeing, employment) but also results in them going over and above their previous state (e.g., increased resilience). This renders PTG an important phenomenon that could be enhanced as part of the support people with cancer receive. IC-Growth has two interconnected paths, namely a research one and another of health policy and best practice recommendations. On the first path, is a sequence of three studies, starting with a systematic review, followed by a cross-sectional study and concludes with a randomized control trial (RCT). The systematic review and close collaboration with experts (e.g., patient associations) will lead to the development of a novel manual to facilitate PTG in groups of people with cancer. The cross-sectional study will explore relationships between variables (e.g., PTG, quality of life, biological variables, illness perceptions, distress, anxiety, depression) in people with cancer (n = 150-180). Lastly, the RCT will evaluate the intervention's effects among three different groups (breast, colorectal, and head and neck cancers, n = 50-60 per group). On the other path, is the development of health policy and best practice recommendations regarding the psychosocial support of people with cancer in Greece. The project's results will be disseminated to stakeholders who provide support to people with cancer (e.g., oncologists, surgeons, psychologists, psychiatrists), through professional associations, a conference on "Psychosocial Support in Oncology", and publications in scientific journals. Overall, IC-Growth is a multidisciplinary project (i.e., psychology, medical, patient organizations, health policy) and joins the clinical, research and policy fields together to workable actions leading to empowering the wider community of people with cancer and improving their care.

DETAILED DESCRIPTION:
Detailed Description IC-Growth is a 24-month, multidisciplinary research and clinical project aimed at enhancing psychosocial care for adults with cancer by promoting post-traumatic growth (PTG)-positive psychological changes following traumatic life crises. While most research emphasizes the negative psychological effects of cancer, IC-Growth focuses on understanding and facilitating PTG as a mechanism to improve well-being, resilience, and quality of life (QoL) beyond pre-diagnosis levels.

The project has two interconnected components:

Research - A sequence of three studies to build, test, and evaluate a novel, manualized PTG intervention for cancer patients:

A systematic review (using PRISMA 2020 and Cochrane standards) to synthesize evidence on PTG interventions.

A cross-sectional study (n = 210-240; breast, colorectal, and head & neck cancer) to examine associations among PTG, QoL, biological markers (e.g., cortisol), illness perceptions, distress, anxiety, and depression.

A randomized controlled trial (RCT) across two centers in Greece (AHEPA University General Hospital and Theageneio Cancer Hospital), comparing a manualized group-based PTG intervention (6-8 weekly sessions, 90 minutes each) with standard care in three cancer populations (70-80 participants per cancer type, randomized into intervention vs. control arms).

Health Policy and Best Practice Development - Using findings from the studies, patient and clinician feedback, and comparisons of national and European oncology guidelines to create evidence-based recommendations for integrating psychosocial interventions into Greek oncology care.

Intervention The PTG intervention will be delivered in groups of 8-10 participants with the same cancer type, facilitated by trained health psychologists. The manual integrates evidence-based therapeutic approaches, including cognitive processing techniques, psychoeducation, cognitive-behavioral elements (e.g., restructuring core beliefs), mindfulness, narrative and existential exercises (e.g., life review, meaning-making), and interpersonal support-building. Sessions are designed to promote growth across PTG's five domains (perception of self, relationships with others, new possibilities, spiritual change, and life appreciation). The intervention's duration is 6-8 weeks, with weekly 90-minute sessions.

Outcomes The primary outcome is PTG, measured via the Post-Traumatic Growth Inventory (PTGI).

Secondary outcomes include:

Quality of life and spiritual well-being (FACIT-Sp and cancer-type specific FACT scales),

Anxiety and depression (Hospital Anxiety and Depression Scale, HADS),

Illness perceptions (Brief Illness Perception Questionnaire, BIPQ),

Distress and trauma impact (Impact of Event Scale-Revised, IES-R),

Biomarkers (cortisol levels as a stress indicator).

Assessments will occur at baseline (pre-intervention) and post-intervention for both control and intervention groups.

Participants Eligible participants are adults (≥18 years) with a diagnosis of breast, colorectal, or head & neck cancer, who have completed planned chemotherapy and hospitalizations, and whose initial diagnosis occurred within the last five years. Exclusion criteria include active psychological or psychiatric treatment, unmanaged mental health conditions, severe cognitive impairment, inability to provide informed consent, non-Greek speakers, cancer relapse(s), diagnosis of another cancer within five years, or life expectancy under one year.

Analysis Statistical analyses will include Pearson and Spearman correlations, factor analysis, network analysis (for cross-sectional findings), and mixed ANOVA/ANCOVA for RCT outcomes. Reliability (Cronbach's alpha) will be assessed for all questionnaires. Qualitative thematic analysis will be used for feedback from participants and professionals to inform feasibility and implementation strategies.

Impact IC-Growth will generate the first manualized PTG intervention in Greece and one of the first RCTs internationally to evaluate PTG across multiple cancer types. Findings will inform the creation of evidence-based best practice and policy recommendations for psychosocial support in oncology care, disseminated via professional associations, a dedicated national conference, and peer-reviewed publications.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years)
2. Having a diagnosis of a. Breast Cancer, b. Colorectal Cancer, or c. Head and Neck Cancer.
3. Having concluded the planned chemotherapy courses and related hospital admissions
4. Having no more than 5 years since the initial diagnosis.

Exclusion Criteria:

1. Being in active psychological or psychiatric treatment
2. Having an unmanaged mental health difficulty
3. Having a severe cognitive impairment
4. Being unable to give informed consent
5. Being unable to speak or read Greek
6. Having one or more relapses
7. Diagnosed with another type of cancer within 5 years prior to recruitment.
8. Having less than one-year life expectancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Growth (PTG) | Baseline and post-intervention (6-8 weeks)
  PTG will be assessed using the Post-Traumatic Growth Inventory (PTGI), a validated 21-item self-report questionnaire measuring positive psychological change following trauma. Higher scores indicate greater post-traumatic growth.

SECONDARY OUTCOMES:
Anxiety and Depression | Measured using the Hospital Anxiety and Depression Scale (HADS), a 14-item validated self-report tool. Higher scores indicate greater levels of anxiety and depression.
  Baseline and post-intervention (6-8 weeks)
Quality of Life and Spiritual Well-being | Baseline and post-intervention (6-8 weeks)
  Measured using the Functional Assessment of Chronic Illness Therapy - Spiritual Well-being (FACIT-Sp) and cancer-type specific scales (e.g., FACT-B, FACT-H&N, FACT-C). Higher scores reflect better perceived quality of life and spiritual well-being.
Distress Related to Traumatic Events | Baseline and post-intervention (6-8 weeks)
  Measured using the Impact of Event Scale-Revised (IES-R), a 22-item self-report instrument assessing subjective distress related to a specific traumatic event. Higher scores indicate greater distress.
Illness Perceptions | Baseline and post-intervention (6-8 weeks)
  Assessed using the Brief Illness Perceptions Questionnaire (BIPQ), which measures cognitive and emotional representations of illness. Higher scores on relevant subscales indicate more negative or threatening illness perceptions.
Salivary Cortisol Levels | Baseline and post-intervention (6-8 weeks)
  Cortisol levels will be measured from saliva samples collected as a biomarker of physiological stress. Lower post-intervention cortisol levels may indicate reduced stress and improved endocrine regulation.

CONTACTS AND LOCATIONS:
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT07108517/Prot_SAP_000.pdf